CLINICAL TRIAL: NCT03137992
Title: A Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Crossover, Multicenter Clinical Study to Assess the Efficacy and Safety of Once Daily Administration of Lupin Tiotropium Bromide Inhalation Powder Compared to SPIRIVA® HANDIHALER® and Placebo in Patients With COPD Including a 12-Week Open Label Extension to Assess Inhaler Robustness
Brief Title: Clinical Endpoint Bioequivalence Study of Test and Reference Inhalation Products in Patients With COPD With Device Robustness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lupin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Lupin Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TB-DPI-301
Record Dates: First submitted 2017-04-30; First posted 2017-05-03 (Actual); Results first posted 2021-04-05 (Actual); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Intervention Model Description: Double-blind, double-dummy, placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Test Product (tiotropium bromide inhalation powder) (Experimental): Once daily administration of test product (tiotropium bromide inhalation powder), 18 mcg for open-label extension (device robustness).
  Interventions: Drug: Test Product (tiotropium bromide inhalation powder)
- Reference Product (Spiriva®) (Active Comparator): Single dose of reference product (Spiriva®) 18 mcg
  Interventions: Drug: Reference Product (Spiriva®)
- Placebo (Placebo Comparator): Single dose of placebo inhalation powder
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Single dose of placebo inhalation powder administered by test and reference dry powder inhalers.
  Arms: Placebo
Drug: Test Product (tiotropium bromide inhalation powder) — Double-Blind: Single dose of test product 18 mcg of test product Open-Label: once daily administration of test product (tiotropium bromide inhalation powder) 18 mcg administered by test dry powder inhaler.
  Arms: Test Product (tiotropium bromide inhalation powder)
Drug: Reference Product (Spiriva®) — Reference product (Spiriva®) 18 mcg.
  Arms: Reference Product (Spiriva®)

SUMMARY:
The purpose of this study is to show bioequivalence of test product to reference product based on baseline-adjusted forced expiratory volume in one second (FEV1).

ELIGIBILITY:
Inclusion Criteria:

* Male and non-pregnant female subjects (40 years of age and older).
* Patients with diagnosis of COPD according to the GOLD guidelines.
* Post-bronchodilator FEV1 <80% of the predicted value at the screening visit.
* Post-bronchodilator FEV1/FVC ratio ≤0.70 at the screening visit.
* Current or former smokers (e.g., with history of = 10 pack-years).
* Written informed consent.

Exclusion Criteria:

* Known respiratory disorder other than COPD including, but not limited to the following: alpha-1 antitrypsin deficiency, cystic fibrosis, significant asthma, active bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, pulmonary edema, or interstitial lung disease.
* History of allergy or hypersensitivity to anticholinergic/muscarinic receptor antagonist agents, beta-2 adrenergic agonists, lactose/milk proteins, or known hypersensitivity to any of the proposed ingredients or components of the delivery system.
* Hospitalization for COPD or pneumonia within 12 weeks prior to the screening visit.
* Treatment for COPD exacerbation within 12 weeks prior to the screening visit.
* Viral or bacterial upper or lower respiratory tract infection, sinusitis, sinus infection, rhinitis, pharyngitis, middle ear infection, urinary tract infection, or illness within 6 weeks prior to the screening visit.
* Abnormal and significant ECG finding prior to the screening, during the run-in and treatment periods.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2018-01-31 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Investigational Research Center Site #1017, Andalusia, Alabama
  - Investigational Research Center Site #1003, Jasper, Alabama
  - Investigational Research Center Site #1008, Glendale, Arizona
  - Investigational Research Center Site #1034, Los Angeles, California
  - Investigational Research Center Site #1028, Riverside, California
  - Investigational Research Center Site #1010, Westminster, California
  - Investigational Research Center Site #1016, Colorado Springs, Colorado
  - Investigational Research Center Site #1026, Clearwater, Florida
  - Investigational Research Center Site #1019, Clearwater, Florida
  - Investigational Research Center Site #1035, Clearwater, Florida
  - Investigational Research Center Site #1036, Orlando, Florida
  - Investigational Research Center Site #1001, North Dartmouth, Massachusetts
  - Investigational Research Center Site #1011, Fridley, Minnesota
  - Investigational Research Center Site #1029, St Louis, Missouri
  - Investigational Research Center Site #1007, Las Vegas, Nevada
  - Investigational Research Center Site #1032, Raleigh, North Carolina
  - Investigational Research Center Site #1037, Columbus, Ohio
  - Investigational Research Center Site #1018, Edmond, Oklahoma
  - Investigational Research Center Site #1009, Oklahoma City, Oklahoma
  - Investigational Research Center Site #1033, Tulsa, Oklahoma
  - Investigational Research Center Site #1005, Medford, Oregon
  - Investigational Research Center Site #1006, Portland, Oregon
  - Investigational Research Center Site #1015, Easley, South Carolina
  - Investigational Research Center Site #1012, Gaffney, South Carolina
  - Investigational Research Center Site #1023, Rock Hill, South Carolina
  - Investigational Research Center Site #1024, Seneca, South Carolina
  - Investigational Research Center Site #1020, Spartanburg, South Carolina
  - Investigational Research Center Site #1025, Spartanburg, South Carolina
  - Investigational Research Center Site #1027, Union, South Carolina
  - Investigational Research Center Site #1004, Knoxville, Tennessee
  - Investigational Research Center Site #1013, El Paso, Texas
  - Investigational Research Center Site #1002, McKinney, Texas
  - Investigational Research Center Site #1030, New Braunfels, Texas
  - Investigational Research Center Site #1031, Newport News, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 377 participants randomized to treatment groups, three subjects did not receive treatment.
Groups:
- Sequence A (T-R-P): Participants received Lupin Tiotropium Bromide Inhalation Powder 18 mcg via LUPINHALER in Period 1 (2 inhalations from one capsule), followed by Spiriva Handihaler 18 mcg in Period 2 (2 inhalations from one capsule), followed by Placebo in period 3 (2 inhalations from one capsule). Select participants who completed Part 1 of the study participated in Part 2 (open-label extension). Subjects received Lupin Tiotropium Bromide Inhalation Powder 18 mcg via LUPINHALER once daily (2 inhalations from one capsule) for 72 days
- Sequence B (R-P-T): Participants received SPIRIVA Handihaler 18 mcg in Period 1 (2 inhalations from one capsule), followed by placebo in Period 2 (2 inhalations from one capsule), followed by Lupin Tiotropium Bromide Inhalation Powder 18 mcg via LUPINHALER in Period 3 (2 inhalations from one capsule). Select participants who completed Part 1 of the study participated in Part 2 (open-label extension). Subjects received Lupin Tiotropium Bromide Inhalation Powder 18 mcg via LUPINHALER once daily (2 inhalations from one capsule) for 72 days
- Sequence C (P-T-R): Participants received Placebo in Period 1 (2 inhalations from one capsule), followed by Lupin Tiotropium Bromide Inhalation Powder 18 mcg via LUPINHALER in Period 2 (2 inhalations from one capsule), followed by SPIRIVA Handihaler 18 mcg in Period 3 (2 inhalations from one capsule). Select participants who completed Part 1 of the study participated in Part 2 (open-label extension). Subjects received Lupin Tiotropium Bromide Inhalation Powder 18 mcg via LUPINHALER once daily (2 inhalations from one capsule) for 72 days
- Sequence D (P-R-T): Participants received Placebo in Period 1 (2 inhalations from one capsule), followed by SPIRIVA Handihaler 18 mcg in Period 2 (2 inhalations from one capsule), followed by Lupin Tiotropium Bromide Inhalation Powder 18 mcg via LUPINHALER in Period 3 (2 inhalations from one capsule). Select participants who completed Part 1 of the study participated in Part 2 (open-label extension). Subjects received Lupin Tiotropium Bromide Inhalation Powder 18 mcg via LUPINHALER once daily (2 inhalations from one capsule) for 72 days
- Sequence E (T-P-R): Participants received Lupin Tiotropium Bromide Inhalation Powder 18 mcg via LUPINHALER in Period 1 (2 inhalations from one capsule), followed by Placebo in Period 2 (2 inhalations from one capsule), followed by SPIRIVA Handihaler 18 mcg in Period 3 (2 inhalations from one capsule). Select participants who completed Part 1 of the study participated in Part 2 (open-label extension). Subjects received Lupin Tiotropium Bromide Inhalation Powder 18 mcg via LUPINHALER once daily (2 inhalations from one capsule) for 72 days
- Sequence F (R-T-P): Participants received SPIRIVA Handihaler 18 mcg in Period 1 (2 inhalations from one capsule), followed by Lupin Tiotropium Bromide Inhalation Powder 18 mcg via LUPINHALER in Period 2 (2 inhalations from one capsule), followed by Placebo in Period 3 (2 inhalations from one capsule). Select participants who completed Part 1 of the study participated in Part 2 (open-label extension). Subjects received Lupin Tiotropium Bromide Inhalation Powder 18 mcg via LUPINHALER once daily (2 inhalations from one capsule) for 72 days
Period: Period 1 (Visit 2)
Arm/Group | Sequence A (T-R-P) | Sequence B (R-P-T) | Sequence C (P-T-R) | Sequence D (P-R-T) | Sequence E (T-P-R) | Sequence F (R-T-P)
Started (Three of the 377 participants enrolled and randomized did not receive any treatment.) | 62 | 63 | 63 | 63 | 62 | 61
Completed (One subject randomized to Sequence A received treatment P in period 1 (visit 2)) | 62 | 63 | 63 | 63 | 62 | 61
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Sequence A (T-R-P) | Sequence B (R-P-T) | Sequence C (P-T-R) | Sequence D (P-R-T) | Sequence E (T-P-R) | Sequence F (R-T-P)
Started | 62 | 63 | 63 | 63 | 62 | 61
Completed | 59 | 59 | 61 | 63 | 60 | 59
Not Completed | 3 | 4 | 2 | 0 | 2 | 2
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Principal Investigator Discretion | 0 | 1 | 0 | 0 | 0 | 0
Not completed — COPD Exacerbation | 1 | 1 | 1 | 0 | 1 | 1
Not completed — Subject Noncompliance | 1 | 0 | 0 | 0 | 1 | 0
Period: Period 2 (Visit 3)
Arm/Group | Sequence A (T-R-P) | Sequence B (R-P-T) | Sequence C (P-T-R) | Sequence D (P-R-T) | Sequence E (T-P-R) | Sequence F (R-T-P)
Started | 59 | 59 | 61 | 63 | 60 | 59
Completed | 56 | 52 | 58 | 58 | 56 | 51
Not Completed | 3 | 7 | 3 | 5 | 4 | 8
Not completed — COPD Exacerbation | 1 | 1 | 0 | 0 | 0 | 1
Not completed — Did not meet continuation criteria | 2 | 3 | 3 | 4 | 3 | 7
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 1 | 0
Period: Washout Period 2
Arm/Group | Sequence A (T-R-P) | Sequence B (R-P-T) | Sequence C (P-T-R) | Sequence D (P-R-T) | Sequence E (T-P-R) | Sequence F (R-T-P)
Started | 56 | 52 | 58 | 58 | 56 | 51
Completed | 54 | 50 | 58 | 57 | 53 | 50
Not Completed | 2 | 2 | 0 | 1 | 3 | 1
Not completed — COPD Exacerbation | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Subject Non-compliance | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 1
Period: Period 3 (Visit 04)
Arm/Group | Sequence A (T-R-P) | Sequence B (R-P-T) | Sequence C (P-T-R) | Sequence D (P-R-T) | Sequence E (T-P-R) | Sequence F (R-T-P)
Started | 54 | 50 | 58 | 57 | 53 | 50
Completed | 48 | 48 | 55 | 57 | 50 | 47
Not Completed | 6 | 2 | 3 | 0 | 3 | 3
Not completed — Did not meet continuation criteria | 6 | 0 | 2 | 0 | 2 | 3
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0 | 1 | 0
Period: Part 2 (Open-label Extension)
Arm/Group | Sequence A (T-R-P) | Sequence B (R-P-T) | Sequence C (P-T-R) | Sequence D (P-R-T) | Sequence E (T-P-R) | Sequence F (R-T-P)
Started (Part 2 of the study enrolled a subset of 125 (from select investigational centers) participants who had successfully completed Part 1 of the study and who met the continuation criteria.) | 22 | 17 | 21 | 25 | 18 | 22
Completed | 20 | 17 | 20 | 24 | 18 | 21
Not Completed | 2 | 0 | 1 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 0
Not completed — COPD exacerbation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Per study team | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Prohibited Medication | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized patients who received a dose of any of the study medications.
Groups:
- Safety Population: The safety analysis population included all patients who received at least one dose of any one of the randomized investigational products and for whom data had been collected after randomization. Patient baseline characteristics are not designated by treatment arms due to the crossover design of the study (treatment groups are not mutually exclusive).
Arm/Group | Safety Population
Number analyzed (Participants) | 374
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 210
  >=65 years | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195
  Male | 179
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 350
  Race: Black/African American | 19
  Race: Asian | 3
  Race: American Indian/Alaska Native | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 7
  Ethnicity: Not Hispanic or Latino | 367
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 374
Baseline Weight [Mean (Standard Deviation); unit: kilograms] | 82.710 (25.452)
Baseline Height [Mean (Standard Deviation); unit: centimeters] | 168.72 (9.927)

OUTCOME MEASURES:

1. Primary Outcome: Baseline Adjusted Mean Change in FEV1 AUC0-24h Post Dose
Description: To show clinical bioequivalence in the efficacy of the test product as a single dose versus reference product based on the baseline adjusted mean change in forced expiratory volume in the first second (FEV1) area under the curve from time zero to 24 hours post dose (AUC0-24h) on day 1 zero to 24 hours post-dose (AUC0-24h). Baseline was defined as the average of the FEV1 values recorded at approximately 30 minutes and 15 minutes before dosing with study medication.
Time Frame: 0-24 hours after dosing on Day 1 of visits 2-4 over a period of approximately 6 weeks
Population: Per-Protocol population
Measure: Least Squares Mean (Standard Error); unit: L*hour
Groups:
- Test Product (Tiotropium Bromide Inhalation Powder): Single dose 18 mcg of test product (tiotropium bromide inhalation powder), a long acting muscarinic receptor antagonist, for double blind portion.
  Once daily administration of test product (tiotropium bromide inhalation powder), 18 mcg for open-label extension (device robustness).
Arm/Group | Test Product (Tiotropium Bromide Inhalation Powder) | Reference Product (Spiriva®)
Number analyzed (Participants) | 291 | 291
L*hour | 2.5644 (0.323) | 2.7370 (0.322)
Statistical Analysis 1: Comparison: Test Product (Tiotropium Bromide Inhalation Powder) vs Reference Product (Spiriva®); A blinded interim analysis was performed after 241 subjects had been randomized with measurable AUC data, which estimated 238 patients would be needed to demonstrate BE with 90% power. Therefore, it was planned that approximately 378 patients would be randomized to allow for a potential 30% loss/withdrawal from the PP population; Test type: Equivalence — Bioequivalence was declared if the 90% CI was entirely contained within the bioequivalence interval, 0.80 to 1.25; Least Squared Mean Ratio = 0.9369, 90% CI 2-sided [0.834 to 1.047] — Fieller's formula was applied to calculate the 90% confidence interval (CI) for the Lupin Tiotropium and Spiriva Handihaler LS mean ratio

2. Primary Outcome: Difference in Baseline Adjusted FEV1 AUC0-24h for Comparison of Lupin Tiotropium Bromide Inhalation Powder (Test) and Spiriva (Reference) to Placebo
Description: This measure is to demonstrate that test product as a single dose and reference product are superior to placebo based on the baseline adjusted mean change in forced expiratory volume in the first second (FEV1) area under the curve from time zero to 24 hours post dose (AUC0-24h) on day 1 zero to 24 hours post-dose (AUC0-24h). Baseline was defined as the average of the FEV1 values recorded at approximately 30 minutes and 15 minutes before dosing with study medication.
Time Frame: 0-24 hours after dosing on Day 1 of visits 2-4 over a period of approximately 6 weeks
Population: Intention-To-Treat population
Measure: Least Squares Mean (Standard Error); unit: L*hour
Arm/Group | Test Product (Tiotropium Bromide Inhalation Powder) | Reference Product (Spiriva®) | Placebo
Number analyzed (Participants) | 372 | 372 | 372
L*hour | 2.90 (0.197) | 3.03 (0.196) | -0.40 (0.199)
Statistical Analysis 1: Comparison: Test Product (Tiotropium Bromide Inhalation Powder) vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — Efficacy of the Test (T) product was demonstrated if the T was shown to be statistically superior to Placebo (p<0.05 [two-tailed]).Outcome variable was Difference in Baseline adjusted FEV1 AUC0-24h; Mixed model repeated measures analysis consisted of effects of treatment, period, and sequence; Least Squared Mean Difference = 3.29, 95% CI 2-sided [2.9386 to 3.646], Standard Error of Mean 0.180
Statistical Analysis 2: Comparison: Reference Product (Spiriva®) vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — Study sensitivity was demonstrated if the Reference (R) product was shown to be statistically superior to Placebo (P) (p <0.05 [two-tailed]). Outcome variable was Difference in Baseline adjusted FEV1 AUC0-24h; Mixed model repeated measures analysis consisted of effects of treatment, period, and sequence; Least Squared Mean Difference = 3.43, 95% CI 2-sided [3.0718 to 3.7797], Standard Error of Mean 0.180

ADVERSE EVENTS:
Time Frame: All AEs/SAEs were assessed through study completion, an average of 14 weeks for participants enrolled in only part 1 of the study and 26 weeks for participants enrolled in part 1 and part 2 of the study. AEs were recorded starting after the patient signed the informed consent form and assessed at each visit.
Description: Adverse events are illnesses or signs/symptoms that appear or worsen during the testing of a drug whether o not considered related to the investigational product (synonyms = medicinal or pharmaceutical product, study medication, clinical trial materials, etc.) including side effects, injury, toxicity, or hypersensitivity reactions. AEs were captured during participant interviews during on-site and telephonic visits.
Groups:
- Test Product (Lupin Tiotropium Bromide Inhalation Powder): Single dose 18 mcg of test product (tiotropium bromide inhalation powder) for double blind portion.
  Once daily administration of test product (tiotropium bromide inhalation powder), 18 mcg for open-label extension (device robustness).
Arm/Group | Test Product (Lupin Tiotropium Bromide Inhalation Powder) | Reference Product (Spiriva®) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/337 | 0/343 | 0/329
Serious Adverse Events (participants affected / at risk) | 0/337 | 0/343 | 0/329
Other Adverse Events (participants affected / at risk) | 0/337 | 0/343 | 0/329

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/92/NCT03137992/SAP_000.pdf
  • Study Protocol (2017-05-11): https://cdn.clinicaltrials.gov/large-docs/92/NCT03137992/Prot_001.pdf